CLINICAL TRIAL: NCT06658587
Title: Clinical Study on the Accuracy of Novel Serological Risk Model in Early Diagnosis of Cholangiocarcinoma Patients
Brief Title: A Novel Serological Risk Model for Early Non-invasive Diagnosis of Cholangiocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-352-01
Record Dates: First submitted 2024-09-11; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Cholangiocarcinoma
Keywords: Hilar Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma; Extrahepatic Cholangiocarcinoma; Early Diagnosis; Non-invasive Diagnosis; Serological; Prognosis; Chemotherapeutic Benefits
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collected blood samples will be tested for the concentration of novel serological markers to construct the serological risk model for differential diagnosis. And the residual samples will be kept in liquid nitrogen for a specific time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University: The cohort of Sun Yat-Sen Memorial Hospital of Sun Yat-sen University is the exploration cohort.
  Interventions: Diagnostic Test: No interventions

INTERVENTIONS:
Diagnostic Test: No interventions — No interventions

SUMMARY:
This is a prospective, observational and exploratory clinical study. The object of this study is to evaluate the accuracy of a novel serological risk model on blood samples in early diagnosis of cholangiocarcinoma patients.

DETAILED DESCRIPTION:
A reliable and accurate preoperative tool capable of early diagnosing malignant cholangiocarcinoma is lacking and urgently needed for clinical practice. This study proposes to establish and evaluate a novel serological risk model on blood samples for non-invasively diagnosing cholangiocarcinoma. The study includes the construction of capable novel serological risk model and the validation of the diagnosis model.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient must sign an informed consent form;
* 2. Age 18-75 years old, both male and female;
* 3. ECOG performance status score (PS score) 0-2;
* 4. Cholangiocarcinoma with resectable tumor lesions;
* 5. Complete the blood collection before treatment;

Exclusion Criteria:

* 1. Accompanied with other primary malignant tumors;
* 2. Patients who have neoadjuvant chemotherapy or other tumor-targeted therapies;
* 3. Incomplete serological examinations or medical history data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had suspected cholangiocarcinoma and completed the blood collection before surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Malignant/Benign status of enrolled suspected cholangiocarcinoma patients by pathological examination | 4 weeks
  The pathological examination results of each enrolled patient will be recorded
Malignant/Benign status of enrolled suspected cholangiocarcinoma patients evaluated by the novel serological risk model | 2 weeks
  The novel serological risk model will be constructed for differential malignant/benign diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PhD, Principal Investigator — Department of Biliary and Pancreatic Surgery, Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No